CLINICAL TRIAL: NCT02159248
Title: 09.017 - A Phase I Study of Tolfenamic Acid With Gemcitabine and Radiation in Patients With Locally Advanced or Metastatic Pancreatic Cancer Requiring Definitive or Palliative Radiation Therapy
Brief Title: Tolfenamic Acid, Gemcitabine and Radiation for Locally Advanced or Metastatic Pancreatic Cancer Requiring Radiation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study closed prior to enrolling any participants.
Sponsor: Orlando Health, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.017
Record Dates: First submitted 2014-06-05; First posted 2014-06-09 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic, gemcitabine, radiation, tolfenamic acid
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tolfenamic acid; Gemcitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolfenamic acid + gemcitabine + radiation (Experimental)
  Interventions: Drug: Tolfenamic acid + gemcitabine + radiation

INTERVENTIONS:
Drug: Tolfenamic acid + gemcitabine + radiation — Cohort 1: 200mg of oral tolfenamic acid, three times per day for 6 1/2 weeks, in combination with weekly intravenous gemcitabine at 400mg/m2 for 5 doses and external beam radiation for 5 1/2 weeks (28 doses at 1.8 Gy/Fx/day).
  Cohort 2: 400mg of oral tolfenamic acid, three times per day for 6 1/2 weeks, in combination with weekly intravenous gemcitabine at 400mg/m2 for 5 doses and external beam radiation for 5 1/2 weeks (28 doses at 1.8 Gy/Fx/day).
  Cohort 3: 600mg of oral tolfenamic acid, three times per day for 6 1/2 weeks, in combination with weekly intravenous gemcitabine at 400mg/m2 for 5 doses and external beam radiation for 5 1/2 weeks (28 doses at 1.8 Gy/Fx/day).
  Cohort 4: 800mg of oral tolfenamic acid, three times per day for 6 1/2 weeks, in combination with weekly intravenous gemcitabine at 400mg/m2 for 5 doses and external beam radiation for 5 1/2 weeks (28 doses at 1.8 Gy/Fx/day).

SUMMARY:
The purposes of this study are to:

* Evaluate the safety and toxicity of tolfenamic acid when used with gemcitabine and radiation therapy in patients with locally advanced or metastatic pancreatic cancer.
* Determine the maximum-tolerated dose (MTD) of tolfenamic acid when used with gemcitabine and radiation in pancreatic cancer.
* Characterize the pharmacokinetic profile of tolfenamic acid when used with gemcitabine and radiation.
* Assess the anti-tumor response to tolfenamic acid when used with gemcitabine and radiation in patients with advanced pancreatic malignancies.

DETAILED DESCRIPTION:
This is a phase I, open-label, non-randomized, single-center, dose-escalation study which utilizes tolfenamic acid in combination with gemcitabine and radiation in patients with locally advanced or metastatic pancreatic malignancies which require definitive or palliative radiation.

Non-steroidal anti-inflammatory drugs (NSAIDs) are known to have a variety of anti-neoplastic mechanisms, including inhibition of cell growth, promotion of apoptosis and inhibition of angiogenesis. Tolfenamic acid is an oral (NSAID) migraine medication which has demonstrated anti-tumor activity in preclinical pancreatic models when used with Gem/XRT (gemcitabine and radiation therapy) and as a single agent.

Each patient enrolled will receive tolfenamic acid in combination with Gem/XRT. Depending on cohort assignment, patients will self-administer tolfenamic acid at either 200mg, 400mg, 600mg or 800mg three times per day. Gemcitabine will be administered intravenously at 400 mg/m2, every seven days for a maximum of 5 doses, starting with the second week of tolfenamic acid administration. Radiation will be given 5 days per week (Monday-Friday) for up to 5 ½ weeks for a maximum dose of 50.4 Gy, beginning with the second week of tolfenamic acid administration.

A maximum of 24 patients will be enrolled in the dose escalation portion of the study. After the maximum tolerated dose (MTD) of tolfenamic acid has been determined, patients will be enrolled in an expansion cohort (at the MTD or the highest dose level achieved if the MTD is not reached) to further assess safety and the anti-tumor response to treatment with tolfenamic acid plus Gem/XRT.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed:

   1. Locally advanced (potentially resectable) pancreatic adenocarcinoma requiring neoadjuvant radiation or
   2. Locally advanced (nonresectable) or metastatic pancreatic adenocarcinoma requiring definitive or palliative radiation therapy
2. Patients may have either measurable or non-measurable disease (according to RECIST criteria, Version 1.1).
3. Age ≥ 18 years
4. ECOG performance status of 0 or 1.
5. A life expectancy of at least 12 weeks.
6. No other concurrent radiotherapy, chemotherapy or immunotherapy.
7. A minimum of 4 weeks must have elapsed since completion of any prior chemotherapy or immunotherapy.
8. Patient must have:

   1. Absolute neutrophil count (ANC) ≥1,000/mm3
   2. Platelets ≥100,000/mm3
   3. Hemoglobin ≥10 g/dL [Transfusion to meet the hemoglobin requirement is acceptable]
   4. Serum creatinine ≤ 1.5 X ULN
   5. Total bilirubin ≤ 1.5 X ULN
   6. Aspartate aminotransferase (AST) ≤ 2.5 X ULN
   7. Alanine aminotransferase (ALT) ≤ 2.5 X ULN
   8. Alkaline phosphatase ≤ 2.5 X ULN
   9. PT/INR ≤ 1.5 X ULN
   10. aPTT ≤ 1.5 X ULN
   11. Urine Protein ≤ Grade 1
9. For patients on warfarin: Must have maintained a stable INR on a stable dose of warfarin for at least 4 weeks prior to start of treatment.

Primary Exclusion Criteria:

1. Patients who have received prior radiation for their current malignancy at the location of interest.
2. Patients who have not recovered (to Grade 1 or less) from adverse events, other than alopecia and neuropathy, caused by previously administered chemotherapeutic agents, at the discretion of the PI/treating physician.
3. Tolfenamic acid use concurrent with, or within 8 weeks prior to the diagnosis of pancreatic cancer.
4. Current use of any non-steroidal anti-inflammatory agents (NSAIDs), including aspirin, (other than tolfenamic acid) within 4 weeks prior to the start of active treatment.
5. Previous history of hypersensitivity reactions (e.g. asthma, rhinitis, angioedema or urticaria) in response to ibuprofen, aspirin or other NSAIDs.
6. History of recurrent peptic ulcer/hemorrhage (two or more distinct episodes).
7. History of gastrointestinal bleeding or perforation related to previous use of NSAIDS.
8. New York Heart Association Functional Classification of 3 or 4.
9. Known autoimmune disease that could preclude the use of radiation, at the discretion of the treating physician.
10. History or evidence of CNS disease (e.g., any brain metastases, primary brain tumor, seizures not controlled with standard medical therapy, or history of stroke).
11. Known HIV positive.
12. Active systemic infection requiring parenteral antibiotic therapy.
13. Receiving systemic steroid therapy. (Inhaled steroid therapy is allowable.)
14. History of other malignancies within the last 5 years with the exception of non- melanoma skin cancer or cervical cancer in situ that has been successfully treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and toxicity | Approximately 16 weeks
  Evaluate the safety and toxicity of escalating doses of tolfenamic acid when used with gemcitabine and radiation in patients with advanced pancreatic malignancies.

SECONDARY OUTCOMES:
Assess the anti-tumor response. | Approximately 16 weeks
  Assess the anti-tumor response to tolfenamic acid when used with gemcitabine and radiation in patients with locally advanced or metastatic pancreatic malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Omar R Kayaleh, M.D., Principal Investigator — Orlando Health
Locations (1):
- UF Health Cancer Center at Orlando Health, Orlando, Florida, United States

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Jutooru I, Chadalapaka G, Abdelrahim M, Basha MR, Samudio I, Konopleva M, Andreeff M, Safe S. Methyl 2-cyano-3,12-dioxooleana-1,9-dien-28-oate decreases specificity protein transcription factors and inhibits pancreatic tumor growth: role of microRNA-27a. Mol Pharmacol. 2010 Aug;78(2):226-36. doi: 10.1124/mol.110.064451. Epub 2010 May 20. PMID 20488920
- [Background] Abdelrahim M, Baker CH, Abbruzzese JL, Safe S. Tolfenamic acid and pancreatic cancer growth, angiogenesis, and Sp protein degradation. J Natl Cancer Inst. 2006 Jun 21;98(12):855-68. doi: 10.1093/jnci/djj232. PMID 16788159
- [Background] Abdelrahim M, Baker CH, Abbruzzese JL, Sheikh-Hamad D, Liu S, Cho SD, Yoon K, Safe S. Regulation of vascular endothelial growth factor receptor-1 expression by specificity proteins 1, 3, and 4 in pancreatic cancer cells. Cancer Res. 2007 Apr 1;67(7):3286-94. doi: 10.1158/0008-5472.CAN-06-3831. PMID 17409437
- [Background] Konduri S, Colon J, Baker CH, Safe S, Abbruzzese JL, Abudayyeh A, Basha MR, Abdelrahim M. Tolfenamic acid enhances pancreatic cancer cell and tumor response to radiation therapy by inhibiting survivin protein expression. Mol Cancer Ther. 2009 Mar;8(3):533-42. doi: 10.1158/1535-7163.MCT-08-0405. Epub 2009 Mar 3. PMID 19258429
- [Background] Maliakal P, Abdelrahim M, Sankpal UT, Maliakal C, Baker CH, Safe S, Herrera LJ, Abudayyeh A, Kaja S, Basha R. Chemopreventive effects of tolfenamic acid against esophageal tumorigenesis in rats. Invest New Drugs. 2012 Jun;30(3):853-61. doi: 10.1007/s10637-010-9622-0. Epub 2011 Jan 4. PMID 21197621
- [Background] Rich TA, Shepard RC, Mosley ST. Four decades of continuing innovation with fluorouracil: current and future approaches to fluorouracil chemoradiation therapy. J Clin Oncol. 2004 Jun 1;22(11):2214-32. doi: 10.1200/JCO.2004.08.009. PMID 15169811
- [Background] A multi-institutional comparative trial of radiation therapy alone and in combination with 5-fluorouracil for locally unresectable pancreatic carcinoma. The Gastrointestinal Tumor Study Group. Ann Surg. 1979 Feb;189(2):205-8. PMID 426553
- [Background] Atasoy BM, Dane F, Ucuncu Kefeli A, Caglar H, Cingi A, Turhal NS, Abacioglu U, Yegen C. Concomitant chemoradiotherapy with low-dose weekly gemcitabine for nonmetastatic unresectable pancreatic cancer. Turk J Gastroenterol. 2011 Feb;22(1):60-4. doi: 10.4318/tjg.2011.0158. PMID 21480113
- [Background] Evans DB, Varadhachary GR, Crane CH, Sun CC, Lee JE, Pisters PW, Vauthey JN, Wang H, Cleary KR, Staerkel GA, Charnsangavej C, Lano EA, Ho L, Lenzi R, Abbruzzese JL, Wolff RA. Preoperative gemcitabine-based chemoradiation for patients with resectable adenocarcinoma of the pancreatic head. J Clin Oncol. 2008 Jul 20;26(21):3496-502. doi: 10.1200/JCO.2007.15.8634. PMID 18640930
- [Background] Joensuu TK, Kiviluoto T, Karkkainen P, Vento P, Kivisaari L, Tenhunen M, Westberg R, Elomaa I. Phase I-II trial of twice-weekly gemcitabine and concomitant irradiation in patients undergoing pancreaticoduodenectomy with extended lymphadenectomy for locally advanced pancreatic cancer. Int J Radiat Oncol Biol Phys. 2004 Oct 1;60(2):444-52. doi: 10.1016/j.ijrobp.2004.03.026. PMID 15380578
- [Background] Moertel CG, Frytak S, Hahn RG, O'Connell MJ, Reitemeier RJ, Rubin J, Schutt AJ, Weiland LH, Childs DS, Holbrook MA, Lavin PT, Livstone E, Spiro H, Knowlton A, Kalser M, Barkin J, Lessner H, Mann-Kaplan R, Ramming K, Douglas HO Jr, Thomas P, Nave H, Bateman J, Lokich J, Brooks J, Chaffey J, Corson JM, Zamcheck N, Novak JW. Therapy of locally unresectable pancreatic carcinoma: a randomized comparison of high dose (6000 rads) radiation alone, moderate dose radiation (4000 rads + 5-fluorouracil), and high dose radiation + 5-fluorouracil: The Gastrointestinal Tumor Study Group. Cancer. 1981 Oct 15;48(8):1705-10. doi: 10.1002/1097-0142(19811015)48:83.0.co;2-4. PMID 7284971
- [Background] Tarnawski AS, Jones MK. Inhibition of angiogenesis by NSAIDs: molecular mechanisms and clinical implications. J Mol Med (Berl). 2003 Oct;81(10):627-36. doi: 10.1007/s00109-003-0479-y. Epub 2003 Sep 6. PMID 13679997
- [Background] Fan F, Wey JS, McCarty MF, Belcheva A, Liu W, Bauer TW, Somcio RJ, Wu Y, Hooper A, Hicklin DJ, Ellis LM. Expression and function of vascular endothelial growth factor receptor-1 on human colorectal cancer cells. Oncogene. 2005 Apr 14;24(16):2647-53. doi: 10.1038/sj.onc.1208246. PMID 15735759
- [Background] Wey JS, Fan F, Gray MJ, Bauer TW, McCarty MF, Somcio R, Liu W, Evans DB, Wu Y, Hicklin DJ, Ellis LM. Vascular endothelial growth factor receptor-1 promotes migration and invasion in pancreatic carcinoma cell lines. Cancer. 2005 Jul 15;104(2):427-38. doi: 10.1002/cncr.21145. PMID 15952180
- [Background] Yang AD, Camp ER, Fan F, Shen L, Gray MJ, Liu W, Somcio R, Bauer TW, Wu Y, Hicklin DJ, Ellis LM. Vascular endothelial growth factor receptor-1 activation mediates epithelial to mesenchymal transition in human pancreatic carcinoma cells. Cancer Res. 2006 Jan 1;66(1):46-51. doi: 10.1158/0008-5472.CAN-05-3086. PMID 16397214
- [Background] Beebe JS, Jani JP, Knauth E, Goodwin P, Higdon C, Rossi AM, Emerson E, Finkelstein M, Floyd E, Harriman S, Atherton J, Hillerman S, Soderstrom C, Kou K, Gant T, Noe MC, Foster B, Rastinejad F, Marx MA, Schaeffer T, Whalen PM, Roberts WG. Pharmacological characterization of CP-547,632, a novel vascular endothelial growth factor receptor-2 tyrosine kinase inhibitor for cancer therapy. Cancer Res. 2003 Nov 1;63(21):7301-9. PMID 14612527
- [Background] Brekken RA, Overholser JP, Stastny VA, Waltenberger J, Minna JD, Thorpe PE. Selective inhibition of vascular endothelial growth factor (VEGF) receptor 2 (KDR/Flk-1) activity by a monoclonal anti-VEGF antibody blocks tumor growth in mice. Cancer Res. 2000 Sep 15;60(18):5117-24. PMID 11016638
- [Background] Cooke SP, Boxer GM, Lawrence L, Pedley RB, Spencer DI, Begent RH, Chester KA. A strategy for antitumor vascular therapy by targeting the vascular endothelial growth factor: receptor complex. Cancer Res. 2001 May 1;61(9):3653-9. PMID 11325835
- [Background] Davis DW, Inoue K, Dinney CP, Hicklin DJ, Abbruzzese JL, McConkey DJ. Regional effects of an antivascular endothelial growth factor receptor monoclonal antibody on receptor phosphorylation and apoptosis in human 253J B-V bladder cancer xenografts. Cancer Res. 2004 Jul 1;64(13):4601-10. doi: 10.1158/0008-5472.CAN-2879-2. PMID 15231672
- [Background] Kozin SV, Boucher Y, Hicklin DJ, Bohlen P, Jain RK, Suit HD. Vascular endothelial growth factor receptor-2-blocking antibody potentiates radiation-induced long-term control of human tumor xenografts. Cancer Res. 2001 Jan 1;61(1):39-44. PMID 11196192
- [Background] Laird AD, Christensen JG, Li G, Carver J, Smith K, Xin X, Moss KG, Louie SG, Mendel DB, Cherrington JM. SU6668 inhibits Flk-1/KDR and PDGFRbeta in vivo, resulting in rapid apoptosis of tumor vasculature and tumor regression in mice. FASEB J. 2002 May;16(7):681-90. doi: 10.1096/fj.01-0700com. PMID 11978732
- [Background] Schlaeppi JM, Wood JM. Targeting vascular endothelial growth factor (VEGF) for anti-tumor therapy, by anti-VEGF neutralizing monoclonal antibodies or by VEGF receptor tyrosine-kinase inhibitors. Cancer Metastasis Rev. 1999;18(4):473-81. doi: 10.1023/a:1006358220123. PMID 10855790
- [Background] Autiero M, Waltenberger J, Communi D, Kranz A, Moons L, Lambrechts D, Kroll J, Plaisance S, De Mol M, Bono F, Kliche S, Fellbrich G, Ballmer-Hofer K, Maglione D, Mayr-Beyrle U, Dewerchin M, Dombrowski S, Stanimirovic D, Van Hummelen P, Dehio C, Hicklin DJ, Persico G, Herbert JM, Communi D, Shibuya M, Collen D, Conway EM, Carmeliet P. Role of PlGF in the intra- and intermolecular cross talk between the VEGF receptors Flt1 and Flk1. Nat Med. 2003 Jul;9(7):936-43. doi: 10.1038/nm884. PMID 12796773
- [Background] Rahimi N, Dayanir V, Lashkari K. Receptor chimeras indicate that the vascular endothelial growth factor receptor-1 (VEGFR-1) modulates mitogenic activity of VEGFR-2 in endothelial cells. J Biol Chem. 2000 Jun 2;275(22):16986-92. doi: 10.1074/jbc.M000528200. PMID 10747927
- [Background] Andre T, Kotelevets L, Vaillant JC, Coudray AM, Weber L, Prevot S, Parc R, Gespach C, Chastre E. Vegf, Vegf-B, Vegf-C and their receptors KDR, FLT-1 and FLT-4 during the neoplastic progression of human colonic mucosa. Int J Cancer. 2000 Apr 15;86(2):174-81. doi: 10.1002/(sici)1097-0215(20000415)86:23.0.co;2-e. PMID 10738243
- [Background] Abdelrahim M, Smith R 3rd, Burghardt R, Safe S. Role of Sp proteins in regulation of vascular endothelial growth factor expression and proliferation of pancreatic cancer cells. Cancer Res. 2004 Sep 15;64(18):6740-9. doi: 10.1158/0008-5472.CAN-04-0713. PMID 15374992
- [Background] Shi Q, Le X, Abbruzzese JL, Peng Z, Qian CN, Tang H, Xiong Q, Wang B, Li XC, Xie K. Constitutive Sp1 activity is essential for differential constitutive expression of vascular endothelial growth factor in human pancreatic adenocarcinoma. Cancer Res. 2001 May 15;61(10):4143-54. PMID 11358838
- [Background] Abdelrahim M, Safe S. Cyclooxygenase-2 inhibitors decrease vascular endothelial growth factor expression in colon cancer cells by enhanced degradation of Sp1 and Sp4 proteins. Mol Pharmacol. 2005 Aug;68(2):317-29. doi: 10.1124/mol.105.011825. Epub 2005 May 9. PMID 15883203
- [Background] Wei D, Wang L, He Y, Xiong HQ, Abbruzzese JL, Xie K. Celecoxib inhibits vascular endothelial growth factor expression in and reduces angiogenesis and metastasis of human pancreatic cancer via suppression of Sp1 transcription factor activity. Cancer Res. 2004 Mar 15;64(6):2030-8. doi: 10.1158/0008-5472.can-03-1945. PMID 15026340
- [Background] Black AR, Black JD, Azizkhan-Clifford J. Sp1 and kruppel-like factor family of transcription factors in cell growth regulation and cancer. J Cell Physiol. 2001 Aug;188(2):143-60. doi: 10.1002/jcp.1111. PMID 11424081
- [Background] Bouwman P, Philipsen S. Regulation of the activity of Sp1-related transcription factors. Mol Cell Endocrinol. 2002 Sep 30;195(1-2):27-38. doi: 10.1016/s0303-7207(02)00221-6. PMID 12354670
- [Background] Safe S, Kim K. Nuclear receptor-mediated transactivation through interaction with Sp proteins. Prog Nucleic Acid Res Mol Biol. 2004;77:1-36. doi: 10.1016/S0079-6603(04)77001-4. No abstract available. PMID 15196889
- [Background] Wang L, Wei D, Huang S, Peng Z, Le X, Wu TT, Yao J, Ajani J, Xie K. Transcription factor Sp1 expression is a significant predictor of survival in human gastric cancer. Clin Cancer Res. 2003 Dec 15;9(17):6371-80. PMID 14695137
- [Background] Yao JC, Wang L, Wei D, Gong W, Hassan M, Wu TT, Mansfield P, Ajani J, Xie K. Association between expression of transcription factor Sp1 and increased vascular endothelial growth factor expression, advanced stage, and poor survival in patients with resected gastric cancer. Clin Cancer Res. 2004 Jun 15;10(12 Pt 1):4109-17. doi: 10.1158/1078-0432.CCR-03-0628. PMID 15217947
- [Background] Corell T. Pharmacology of tolfenamic acid. Pharmacol Toxicol. 1994;75 Suppl 2:14-21. doi: 10.1111/j.1600-0773.1994.tb01991.x. No abstract available. PMID 7816775
- [Background] Pedersen SB. Biopharmaceutical aspects of tolfenamic acid. Pharmacol Toxicol. 1994;75 Suppl 2:22-32. doi: 10.1111/j.1600-0773.1994.tb01992.x. PMID 7816776
- [Background] Pentikainen PJ, Penttila A, Neuvonen PJ, Khalifah RG, Hignite CE. Human metabolism of tolfenamic acid. I. Isolation, preliminary characterization and pharmacokinetics of tolfenamic acid and its metabolites. Eur J Drug Metab Pharmacokinet. 1982 Oct-Dec;7(4):259-67. doi: 10.1007/BF03189628. No abstract available. PMID 7166178
- [Background] Rozencweig M, Von Hoff DD, Staquet MJ, Schein PS, Penta JS, Goldin A, Muggia FM, Freireich EJ, DeVita VT Jr. Animal toxicology for early clinical trials with anticancer agents. Cancer Clin Trials. 1981;4(1):21-8. PMID 6783332